CLINICAL TRIAL: NCT05662852
Title: A Clinical Study of the Safety and Antibody Responses of Plasma Donors Vaccinated With a Licensed Tdap Vaccine for a Hyperimmunization Program
Brief Title: Safety and Immunogenicity Study of Tdap Vaccinations for Plasma Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ABO Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ABO-TET-01
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Tetanus, Diphtheria and Acellular Pertussis Vaccination
Keywords: Plasma; Plasma Donor; Plasma Donation; Hyperimmunization; Tetanus; Immunoglobulin
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tdap for Plasma Donors (Experimental): Dose: 0.5 mL; Route: Intramuscular (IM) in the deltoid muscle; Frequency: Every 90 days; Duration: 5 doses over 1 year.
  Interventions: Biological: Tdap

INTERVENTIONS:
Biological: Tdap — Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed Suspension manufactured by Sanofi Pasteur
  Other Names: Adacel

SUMMARY:
The goal of this clinical trial is to investigate the safety and tetanus antibody response to a Tdap vaccine in healthy plasma donors. The main question it aims to answer are:

* Is it safe to give this vaccine multiple times over one year to plasma donors since the package insert for this vaccine indicates that it should administered once every 10 years?
* What is the tetanus antibody response over time in these donors after receiving the vaccine multiple times during the study?

Participants will receive a Tdap vaccination every 3 months ±2 weeks for 12 months (5 vaccinations) with a 6 month follow-up after the last vaccination. After obtaining informed consent and screening for eligibility including plasmapheresis donor eligibility, subjects will have other baseline assessments performed and if eligible, will receive the scheduled vaccinations, will be assessed for adverse events (AEs) and have plasma samples collected for antibody titers each month thereafter for 11 months, and then at 1 and 6 months after the last vaccination. As these subjects are participating in a standard donor plasmapheresis donor program, assessments for donor eligibility and routine plasmapheresis will be performed; however, only the data specifically required to meet the objectives of this study will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 to 63 years
* Females of childbearing potential who agree to employ highly effective birth control measures during the study
* Signed the informed consent form (ICF)
* Met all of the criteria required to be a Normal Source Plasma donor
* Subject is not participating in any other immunization program
* Subject has not had a Tdap vaccination in the last 90 days before the first study vaccination

Exclusion Criteria:

* Subject is pregnant
* Subject has a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data
* Subject has repeated reactions or hypersensitivity to components in the vaccine
* Subject has history of a severe reaction to any immunization
* Subject has a history of Guillain-Barré Syndrome
* The Investigator concludes that the anticipated vaccination site (deltoid area) is not suitable for AE assessment

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 18 months
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as an adverse event occurring after first study treatment. A serious TEAE was defined as an AE that resulted in any of the following outcomes: death; life-threatening; inpatient hospitalization or prolongation of hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, an important medical event that based on appropriate medical judgment may jeopardize the subject and may require medical or surgical intervention to prevent one of the aforementioned outcomes.

SECONDARY OUTCOMES:
Anti-tetanus Antibody Titers in Participants Over Time | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 18
  Anti-tetanus antibody titer levels after each vaccination presented at geometric means (GeoMean) over time.
Number of Participants With Post Vaccination Anti-tetanus Antibody Range Levels | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 18
  The numbers and percentages of participants whose post vaccination antibody levels were <5 IU/mL; ≥5 IU/mL to 10 IU/mL; >10 IU/mL to 15 IU/mL; and, >15 IU/mL after each vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Thaler, DO, Principal Investigator — Center Medical Director
Locations (1):
- ABO Plasma, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No